CLINICAL TRIAL: NCT07331259
Title: C3 Glomerulopathy Patient Characteristics and Treatment Response to Iptacopan in Routine Care: Analysis of Medical Charts (CHART-C3G)
Brief Title: CHART-C3G/CLNP023B12011
Status: Not yet recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023B12011
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: C3 Glomerulopathy; Complement-mediated Kidney Disease; Proteinuria
Keywords: NIS-PDC; Germany; C3G; Iptacopan; estimated Glomerular Filtration Rate
MeSH Terms: conditions — Proteinuria | interventions — iptacopan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Iptacopan: Adult patients with C3G initiating iptacopan treatment in routine care
  Interventions: Other: Iptacopan

INTERVENTIONS:
Other: Iptacopan — There is no treatment allocation for NIS trials. Patients administered Iptacopan by prescription will be enrolled.
  Other Names: LNP023B

SUMMARY:
This is a non-interventional chart abstraction cohort study with longitudinal follow up. Patients with C3G treated with iptacopan will be enrolled and characterized (i.e., systematically describe and summarize) regarding their medical history and iptacopan use and evaluated for clinical events, outcomes, and laboratory measurements upon and after iptacopan treatment initiation. Medical charts will be used to obtain secondary pseudonymized patient-level data with reference to 2 time anchors: at index date (date of iptacopan treatment initiation) with baseline covering 12 months prior to index date, and at 12-month follow-up (twelve months after the index date).The observation period includes baseline plus follow-up.

Iptacopan will be used as prescribed by the clinician in accordance with the terms of the marketing authorization. This Novartis-sponsored study, mainly executed by a contract research organization (CRO), will use secondary data from EHR obtained through reference centers/ centers of excellence in glomerular diseases in Germany.

The primary objective of this study is to characterize the demographic and clinical profiles of adult patients diagnosed with C3G upon iptacopan treatment initiation.

DETAILED DESCRIPTION:
Until recently, there are no approved disease-specific treatments for C3G, although there is significant interest in the therapeutic potential of complement inhibition.

Iptacopan, the first oral effective targeted disease-modifying proximal complement inhibitor developed by Novartis, has been approved in April 2025 for the treatment of adults with C3G.

The primary objective of this study is to characterize the demographic and clinical profiles of adult patients diagnosed with C3G upon iptacopan treatment initiation.

By analyzing key endpoints such as age, sex, ethnicity, BMI, clinical symptoms, proteinuria, blood pressure, serum creatinine, eGFR, serum C3 levels, and renal histological parameters, we aim to better understand disease progression and treatment outcomes.

Additionally, we will assess CKD stages, history of kidney failure, dialysis status, transplant status, and comorbidities to identify the characteristics of patients treated with iptacopan.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of C3G (confirmed by biopsy, only if available)
* Aged ≥18 years at time of index date.
* At least 6 months of baseline period preceding index date.
* Users of iptacopan treatment including those who have discontinued iptacopan within the last twelve weeks.

Exclusion Criteria:

* Interventional C3G clinical trial participation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years clinically diagnosed with C3G from participating study sites who initiate iptacopan during the period between 31-Mar-2025 and 31-Dec-2025
Sampling Method: Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Demographics: Number of patients by age | Baseline
  Age at baseline in years
Demographics: Number of patients by sex | Baseline
  Female Male
Demographics: Number of patients by site | Baseline
  Academic hospital Other sites
Demographics: Body mass index | Baseline
  Body mass index reported at baseline, or the closest value before baseline. In the absence of records for body mass index, it can be calculated using records of height and weight.
Demographics: Number of patinets with Biopsy confirming C3G | Baseline
  No Yes
Clinical symptoms: Proteinuria - Number of participants by 24-hour uPCR | Baseline
  No Yes 24-hour uPCR < 1 g/g 24-hour uPCR ≥ 1 g/g
Proteinuria - Number of participants by spot uPCR | Baseline
  No Yes Spot uPCR < 1 g/g Spot uPCR ≥ 1 g/g
Proteinuria, 24-hour uPCR in g/g | Baseline
  Absolute value of uPCR based on a 24-hour urine collection
Proteinuria, spot uPCR in g/g | Baseline
  Absolute value of uPCR based on a spot urine collection
Clinical symptoms: Albuminuria | Baseline
  No Yes
Albuminuria - Number of participants by spot uACR | Baseline
  No Yes
Albuminuria, 24-hour uACR in g/g | Baseline
  Absolute value of uACR based on a 24-hour urine collection
Albuminuria, spot uACR in g/g | Baseline
  No Yes
Clinical symptoms: Number of participants by Hematuria - dipstick results | Baseline
  No Yes Microscopic (≥3RBCs/HPF) Macroscopic (visible to the naked eye)
Hematuria - Number of participants by urinalysis results | Baseline
  0-2 red blood cells
  ≥3 red blood cells
Hematuria - urinalysis, number of red blood cells | Baseline
  Number of red blood cells detected through urinalysis
Clinical symptoms: Number of participants with presence of edema | Baseline
  Presence of edema. No Yes
Clinical symptoms: Systolic and diastolic blood pressure | Baseline
  Blood pressure measurement
Clinical symptoms: Number of participants with hypertension | Baseline
  Defined as systolic blood pressure ≥140 mmHg or a diastolic blood pressure ≥90 mmHg No Yes
Clinical symptoms: Serum creatinine at baseline | Baseline
  Absolute value of serum creatinine
Clinical symptoms: Reported eGFR at baseline | Baseline
  Based on medical records of eGFR
Clinical symptoms: Number of participants by equation used in reported eGFR at baseline | Baseline
  2021 CKD-EPI creatinine 2021 CKD-EPI creatinine-cystatin C 2012 CKD-EPI cystatin C 2012 CKD-EPI creatinine-cystatin C 2009 CKD-EPI creatinine MDRD (based on creatinine) Cockroft-Gault (based on creatinine) Schwartz equation (based on creatinine) Not specified
Clinical symptoms: Computed eGFR at baseline | Baseline
  eGFR computed in the study analysis
Clinical symptoms: Serum C3 at baseline | Baseline
  Reference range: LLN = 4.33-5.00 μmol/L ULN = 9.05-11.16 μmol/L
Clinical events and outcomes: Time since C3G diagnosis (days/months) | Baseline
  Time since the first C3G diagnosis to baseline
Clinical events and outcomes: Number of participants with Chronic Kidney Disease (CKD) and stage | Baseline
  No Yes Stage 1 Stage 2 Stage 3 Stage 4 Stage 5
Clinical events and outcomes: Number of participants with history of kidney failure | Baseline
  No Yes (either of the categories below) eGFR ≤ 15 History of dialysis History of kidney transplant
Clinical events and outcomes: Number of participants by dialysis status | Baseline
  No Yes Dialysis at diagnosis of C3G Maintenance dialysis Other types
Clinical events and outcomes: Time from C3G diagnosis to dialysis (months) | Baseline
  Concerns only patients with dialysis at or before baseline
Clinical events and outcomes: Time from dialysis to baseline (months) | Baseline
  Concerns only patients with dialysis at or before baseline
Clinical events and outcomes: Number of participants by transplant status at baseline | Baseline
  No (native kidney) Yes Biopsy-confirmed disease in native kidney No evidence of disease recurrence Recurrent disease in transplanted kidney
Clinical events and outcomes: Time from C3G diagnosis to kidney transplant before baseline (months) | Baseline
  Concerns only patients with a kidney transplant (or kidney transplant failure) at or before baseline
Clinical events and outcomes: Time from kidney transplant before baseline to baseline (months) | Baseline
  Concerns only patients with a kidney transplant (or kidney transplant failure) at or before baseline
Clinical events and outcomes: Number of participants with C3G disease recurrence post-transplant and/or transplant failure | Baseline
  Concerns only patients with a kidney transplant (or kidney transplant failure) at or before baseline.
  No Yes
Clinical events and outcomes: Number of participants with comorbidities | Baseline
  For example, history of heart failure, history of stroke, diabetes mellitus, dementia, malignancy
Renal histopathological parameters: Number of participants with presence of cysts | Baseline
  No Yes
Renal histopathological parameters: Number of participants with presence of tumors | Baseline
  No Yes
Renal histopathological parameters: Number of participants with presence of interstitial fibrosis or tubular atrophy | Baseline
  Mild Moderate Severe
Renal histopathological parameters: Number of participants with presence of glomerulosclerosis | Baseline
  Mild Moderate Severe
Renal histopathological parameters: Endocapillary hypercellularity | Baseline
  Presence of cells in capillary loops with loop occlusion 0 = 0% (Essentially normal or no lesion)
  1. = 1-25% (Only a small fraction of loops are occluded by hypercellularity)
  2. = 26-50% (About one-quarter to half of the loops show occlusion)
  3. = ≥51% (More than half of the loops are occluded, indicating extensive endocapillary proliferation)
Renal histopathological parameters: Neutrophils in capillary lumens (each glomerulus is scored) | Baseline
  0 = 0% (No neutrophils in any capillary loops of the glomerulus)
  1. = 1-25% (Mild involvement: neutrophils present in up to ¼ of loops)
  2. = 26-50% (Moderate involvement: neutrophils in about ¼ to half of loops)
  3. = ≥51% (Severe involvement: neutrophils in more than half of loops)
Renal histopathological parameters: Mesangial hypercellularity | Baseline
  More than 4 cells in a mesangial area away from the hilum
  0 = 0% (No mesangial areas with >4 cells)
  1. = 1-25% (Mild involvement: 1-25% of mesangial areas show hypercellularity)
  2. = 26-50% (Moderate involvement: 26-50% of mesangial areas affected)
  3. = ≥51% (Severe involvement: More than half of mesangial areas show hypercellularity)
Renal histopathological parameters: Necrosis | Baseline
  Necrosis in glomerular pathology refers to active destructive lesions characterized by:
  Disruption of the glomerular basement membrane (GBM) Fibrin exudation into Bowman's space or capillary loops Karyorrhexis (fragmentation of nuclei of inflammatory cells) - at least 2 of these 3 lesions need to be present to meet the criteria for necrosis.
  0 = 0% (No glomeruli show necrosis)
  1. = 1-10% (Mild: 1-10% of glomeruli have necrosis)
  2. = 11-25% (Moderate: 11-25% of glomeruli affected)
  3. = ≥25% (Severe: More than 25% of glomeruli show necrosis)
Renal histopathological parameters: Cellular or fibrocellular crescents | Baseline
  0 = 0% (No crescents in any glomeruli)
  1. = 1-10% (Mild: 1-10% of glomeruli have crescents)
  2. = 11-25% (Moderate: 11-25% of glomeruli affected)
  3. = >25% (Severe: More than 25% of glomeruli show crescents)
Renal histopathological parameters: Activity index | Baseline
  A score between 0 and 15, calculated by summing up the scores from the activity index parameters above (Endocapillary hypercellularity,. Neutrophils in capillary lumens, Mesangial hypercellularity, Necrosis and Cellular or fibrocellular crescents).
  Score 0: No active lesions. The kidney shows chronic changes only, but no ongoing inflammation.
  Higher score implies not aggressively active, and kidney damage is likely stable or progressing slowly.
Renal histopathological parameters: score inflammation assessment scale | Baseline
  Both continuous (score inflammation assessment scale) and categorically (none, mild, moderate, severe).
  Continuous Scale (Numeric Score)
  1. Low score (e.g., 0-3) Minimal inflammatory activity
  2. High score (e.g., ≥9) Extensive active lesions (necrosis, crescents, heavy infiltration)
  Categorical Scale (None, Mild, Moderate, Severe)
  1. None: No significant inflammation; likely chronic or inactive disease.
  2. Mild: Small, focal involvement; early or controlled disease.
  3. Moderate: Widespread but not diffuse; active disease needing treatment.
  4. Severe: Diffuse, aggressive inflammation; high risk of rapid progression to renal failure.
Renal histopathological parameters: Number of participants by typo of inflammation | Baseline
  Type of inflammation: none, mild, moderate, severe
Chronicity index parameters: Number of participants with glomerular (or segmental) sclerosis | Baseline
  0 = ≤10%
  1. = 11-25%
  2. = 26-50%
  3. = ≥51%
Chronicity index parameters: Number of participants with Fibrous crescents | Baseline
  0 = none
  1. = ≤25%
  2. = 26-50% 3= >51%
Chronicity index parameters: Number of participants with tubular atrophy | Baseline
  0 = ≤5%
  1. = 6-25%
  2. = 26-50%
  3. = ≥51%
Chronicity index parameters: Number of participants with interstitial fibrosis | Baseline
  0 = ≤5%
  1. = 6-25%
  2. = 26-50%
  3. = ≥51%
Renal histopathological parameters: Chronicity index | Baseline
  A score between 0 and 12, calculated by summing up the scores from the chronicity index parameters above (Glomerular (or segmental) sclerosis, Fibrous crescents, Tubular atrophy and Interstitial fibrosis)
  Lower scores indicate less chronic damage, higher scores indicate more scarring and poor prognosis.
  0-3 (Minimal to Mild)
  → Very little irreversible damage. Prognosis is generally favorable if activity index is also low.
  4-6 (Moderate)
  * Significant chronic changes; recovery potential is limited. 7-12 (Severe)
  * Extensive scarring; immunosuppression unlikely to reverse damage

SECONDARY OUTCOMES:
Clinical events and outcomes: Number of participants with kindney failure during follow-up | Up to 12 months
  No Yes
Clinical events and outcomes: Time from C3G diagnosis to kidney failure and time from baseline to kidney failure | Up to 12 months
  Concerns only patients with kidney failure during follow-up
Clinical events and outcomes: Number of participants with dialysis during follow-up | Up to 12 months
  No Yes Maintenance dialysis Other types
Clinical events and outcomes:Time from kidney failure to first dialysis (months) | Up to 12 months
  Concerns only patients with dialysis during follow-up
Clinical events and outcomes: Time from baseline to first dialysis (months) | Up to 12 months
  Concerns only patients with dialysis during follow-up
Clinical events and outcomes: Time from kidney failure to maintenance dialysis (months) | Up to 12 months
  Concerns only patients with maintenance dialysis during follow-up
Clinical events and outcomes: Time from C3G diagnosis to maintenance dialysis (months) | Up to 12 months
  Concerns only patients with maintenance dialysis during follow-up
Clinical events and outcomes: Time from baseline to maintenance dialysis (months) | Up to 12 months
  Concerns only patients with maintenance dialysis during follow-up
Clinical events and outcomes: Number of participants with complete remission (controlled) of C3G during follow-up | Up to 12 months
  No Yes
Clinical events and outcomes: Number of participants with nephrotic-range and non-nephrotic range proteinuria during follow-up | Up to 12 months
  Non-nephrotic-range proteinuria (0.15-3.5 g of protein in a 24-hour urine collection) Nephrotic-range proteinuria (> 3.5 g of protein in a 24- hour urine collection)
Clinical events and outcomes: Number of participants with renal relapse, progression to a higher CKD stage, or chronic renal replacement therapy during follow-up | Up to 12 months
  No Yes Renal relapse Progression to a higher CKD stage Chronic renal replacement therapy
Clinical events and outcomes: Number of transplant failures per patient during follow-up | Up to 12 months
  Transplant failure is defined as a follow-up record of either maintenance dialysis, sustained eGFR <15 mL/min/1.73m², or re-transplant
Clinical events and outcomes: Number of participants with CKD and stage at 12-month follow-up | Up to 12 months
  No Yes Stage 1 Stage 2 Stage 3 Stage 4 Stage 5
Clinical events and outcomes: Number of participants by transplant status at 12-month follow-up | Up to 12 months
  No (native kidney) Yes Biopsy-confirmed disease in native kidney No evidence of disease recurrence Recurrent disease in transplanted kidney
Clinical events and outcomes: Number of participants with Kidney transplant during follow-up | Up to 12 months
  No Yes No transplant failure during follow-up Transplant failure during follow-up
Clinical events and outcomes: Time from kidney failure to transplant during follow-up (months) | Up to 12 months
  Concerns only patients with a kidney transplant (or kidney transplant failure) during follow-up
Clinical events and outcomes: Time from transplant during follow-up to post- transplant C3G disease recurrence (months) | Up to 12 months
  Concerns only patients with a kidney transplant (or kidney transplant failure) during follow-up and a post-transplant C3G disease recurrence during follow-up
Clinical events and outcomes: Time from transplant to transplant failure (months) | Up to 12 months
  Concerns only patients with a kidney transplant during follow-up and a transplant failure during follow-up
Clinical events and outcomes: Number of participants with C3G disease recurrence post-transplant and/or transplant failure | Up to 12 months
  Concerns only patients with a kidney transplant (or kidney transplant failure) during follow-up.
  No Yes C3G disease recurrence post-transplant Transplant failure C3G disease recurrence post-transplant and transplant failure
Clinical events and outcomes: Time from C3G disease recurrence to transplant failure | Up to 12 months
  Concerns only patients with the combination of kidney transplant during follow-up, C3G disease recurrence post-transplant, and subsequent transplant failure
Clinical events and outcomes: Time from transplant at any time to post- transplant C3G disease recurrence | Up to 12 months
  Concerns patients with a kidney transplant (or kidney failure) at any time, including baseline and follow-up, and post-transplant C3G disease recurrence at any time, including baseline and follow-up
Clinical events and outcomes: Number of participants with death during follow-up | Up to 12 months
  No Yes
Clinical events and outcomes: Number of participants by cause of Death | Up to 12 Months
  Concerns only patients with death during follow-up. Kidney failure Infectious disease Cardiovascular disease Other causes
Laboratory measurements: Serum creatinine or eGFR | 6 months, 12 months and 24 months before baseline and up to 12 months follow-up
  Serum creatinine (preferred) or eGFR
Laboratory measurements: eGFR slope during the 24months prior to baseline | 24 months prior to baseline and 12 months post baseline
  Average eGFR slope computed using baseline computed eGFR and available historical serum creatinine values (preferred) or eGFR
Laboratory measurements: Change in reported eGFR from baseline to 12-month follow-up, mL/min/1.73m | Baseline, Month 12
  Difference in absolute value of reported eGFR between end of follow-up and baseline
Laboratory measurements: Equation used in reported 12-month follow-up eGFR | Month 12 follow-up
  Equation used in reported 12-month follow-up eGFR:
  2021 CKD-EPI creatinine 2021 CKD-EPI creatinine-cystatin C 2012 CKD-EPI cystatin C MDRD (based on creatinine) Cockroft-Gault (based on creatinine) Schwartz equation (based on creatinine) Not specified
Laboratory measurements: Follow-up serum creatinine or eGFR 6 months after baseline | Up to 12 months
  Serum creatinine (preferred) or eGFR at 6 months after baseline
Laboratory measurements: eGFR slope during the 12 months after baseline, mL/min/1.73m²/year | Up to 12 months
  Average eGFR slope computed using available follow-up serum creatinine values (preferred) or eGFR
Laboratory measurements: Change in computed eGFR from baseline to 12-month, mL/min/1.73m | Baseline, Month 12
  Difference in absolute value of computed eGFR between end of follow-up and baseline
Laboratory measurements: Number of participants with Proteinuria 24-hour uPCR | Up to 12 months
  No Yes 24-hour uPCR < 1 g/g 24-hour uPCR ≥ 1 g/g
Laboratory measurements: Number of participants with Proteinuria at 12-month follow-up - spot uPCR | Up to 12 months
  No Yes Spot uPCR < 1 g/g Spot uPCR ≥ 1 g/g
Laboratory measurements: Proteinuria at 12-month, spot uPCR in g/g | Up to 12 months
  Absolute value of uPCR based on a spot urine collection
Laboratory measurements: Proteinuria at 12-month follow-up, 24-hour uPCR in g/g | Up to 12 months
  Absolute value of uPCR based on a 24-hour urine collection
Laboratory measurements: Change in proteinuria from baseline to 12-month follow-up, 24-hour uPCR in g/g | Baseline, Month 12
  Difference in absolute value of 24-hour uPCR from baseline to 12-month follow-up, in g/g
Laboratory measurements: Change in proteinuria from baseline to 12-month follow-up, spot uPCR in g/g | Baseline, Month 12
  Difference in absolute value of spot uPCR from baseline to 12-month follow-up, in g/g
Laboratory measurements: Change in proteinuria from baseline to 12-month follow-up in mg/mmol - 24-hour uPCR | Baseline, Month 12
  Change of uPCR based on a 24-hour urine collection from baseline to 12-month follow-up, in mg/mmol Below 100 mg/mmol Above 100 mg/mmol
Laboratory measurements: Change in proteinuria from baseline to 12-month follow-up in mg/mmol - spot uPCR | Baseline, Month 12
  Change of uPCR based on a spot urine collection from baseline to 12-month follow-up, in mg/mmol Below 100 mg/mmol Above 100 mg/mmol
Laboratory measurements: Change in proteinuria from baseline to 12-month follow-up in g/g - 24-hour uPCR | Baseline, Month 12
  Change of uPCR based on a 24-hour urine collection from baseline to 12-month follow-up, in mg/mmol Below 1 g/g Above 1 g/g
Laboratory measurements: Change in proteinuria from baseline to 12-month follow-up in g/g - spot uPCR | Baseline, Month 12
  Change of uPCR based on a spot urine collection from baseline to 12-month follow-up, in mg/mmol Below 1 g/g Above 1 g/g
Laboratory measurements: Number of participants with albuminuria | Up to 12 months
  No Yes
Laboratory measurements: Number of participants with Albuminuria at 12-month follow-up - spot uACR | Up to 12 months
  No Yes
Laboratory measurements: Albuminuria at 12-month follow-up, 24-hour uACR in g/g | Up to 12 months
  Absolute value of uACR based on a 24-hour urine collection
Laboratory measurements: Albuminuria at 12-month follow-up, spot uACR in g/g | Up to 12 months
  Absolute value of uACR based on a spot urine collection
Laboratory measurements: Change in albuminuria from baseline to 12-month follow-up, 24-hour uACR in g/g | Baseline, Month 12
  Difference in absolute value of 24-hour uACR from baseline to 12-month follow-up
Laboratory measurements: Change in albuminuria from baseline to 12-month follow-up, spot uACR in g/g | Baseline, Month 12
  Difference in absolute value of spot uACR from baseline to 12-month follow-up
Laboratory measurements: Number of participants with Hematuria dipstick | Up to 12 months
  No Yes Microscopic Macroscopic
Laboratory measurements: Hematuria - Number of participants by urinalysis results | Up to 12 months
  0-2 red blood cells
  ≥3 red blood cells
Laboratory measurements: Hematuria - urinalysis, number of red blood cells | Up to 12 months
  Number of red blood cells detected through urinalysis
Laboratory measurements: Change in hematuria from baseline to 12-month follow-up | Baseline, Month 12
  No change From no to yes From yes to no
Laboratory measurements: Change in hematuria on urinalysis from baseline to 12-month follow-up, number of red blood cells | Baseline, Month 12
  Difference in absolute number of red blood cells detected through urinalysis from baseline to 12-month follow-up
Laboratory measurements: Number of participants with presence of autoantibodies | Up to month 12 follow-up
  No Presence of any of the below autoantibodies C3NeF C4NeF C5NeF Anti-factor H autoantibodies Anti-factor B autoantibodies Anti-C3b autoantibodies
Laboratory measurements: CH50 and CH100 | Up to month 12 follow up
  CH50: The 50% activity of the classic pathway of the complement CH100: Total activity of the classic pathway of the complement
Laboratory measurements: AH50 and AH100 | Up to month 12 follow-up
  AH50: The 50% activity of the alternative pathway of the complement AH100: Total activity of the alternative pathway of the complement
Laboratory measurements: Wieslab activity of the alternative pathway of complement | Up to month 12 follow-up
  Wieslab activity values are provided on a scale such that 100% of activity is normal activity. Full inhibition of alternative pathway corresponds to a value of 0
Laboratory measurements: Serum C3, Serum C4 and Serum C5 | Up to month 12 follow-up
  Serum C3 Reference range: LLN = 4.33-5.00 µmol/L ; ULN = 9.05-11.16 µmol/L Serum C4 Reference range: LLN = 0.50-0.70 µmol/L ; ULN = 2.00-2.60 µmol/L Serum C5 Reference range: LLN = 50 µg/mL ; ULN = 115 µg/mL
Laboratory measurements: Fibrinogen Degradation; (FD) | Up to month 12 follow-up
  Reference range:
  LLN = 1437 µg/L ULN = 3966 µg/L
Laboratory measurements: fragment a of complement factor B (Ba) | Up to month 12 follow-up
  Reference range:
  LLN = 338 ng/mL ULN = 1164 ng/mL
Laboratory measurements: fragment b of complement factor B (Bb) | Up to 12 months follow-up
  Reference range:
  LLN = 0.49 mg/L ULN = 1.42 mg/L
Laboratory measurements: soluble terminal complement activation fragment (sC5b-9) | Up to 12 months follow-up
  Reference range: LLN = 95 µg/L ULN = 467 µg/L
Disease management: Number of participants by status of vaccination and prophylactic antibiotic at baseline | Up to 12 months follow up
  Vaccination status at baseline Neisseria meningitidis Staphylococcus pneumoniae Vaccinated for both Received prophylactic antibiotic treatment
Disease management: Number of participants by Iptacopan daily dose | Baseline and up to 12 months follow-up
  Iptacopan daily dose at initiation and at the end of follow-up (or at discontinuation)
Disease management: Number of participants by Iptacopan daily dose change from baseline to the end of follow-up | Baseline, up to month 12 follow-up
  Dose increase Dose decrease No modification
Disease management: Time to first modification of iptacopan dosage (days) | Up to 12 months-follow up
  Time from baseline to the first modification of the daily dose of iptacopan
Disease management: Number of participants by reason of modification of iptacopan dosage during follow-up | Up to 12 months follow-up
  Reason of modification of iptacopan dosage during follow-up
Disease management: Missed or delayed dose of iptacopan during follow-up | Up to 12 months follow-up
  0 1-2 3-4 5 or more
Disease management: Number of participants with prior use of immunosuppressive medication | Up to month 12 follow-up
  Immunosuppressive medication used before baseline and/or discontinued before baseline.
  No Yes Corticosteroids Prednisolone Methylprednisolone Cyclophosphamide Complement inhibitors C5 inhibitors (e.g., eculizumab) Other complement inhibitors (specify) Mycophenolate mofetil Rituximab Tacrolimus mTORi (everolimus/sirolimus) Other C3G medication (specify)
Disease management: Time from C3G diagnosis to the first complement inhibitor before baseline | Baseline
  Concerns only patients with prior use of complement inhibitors.
Disease management: Number of participants by concomitant C3G treatments | Up to 12 months follow-up
  Use of other C3G treatment in concomitance to iptacopan. No Yes ACEi/ARB Corticosteroids Prednisolone Methylprednisolone Cyclophosphamide Complement inhibitors C5 inhibitors (e.g., eculizumab) Other complement inhibitors (specify) Mycophenolate mofetil Rituximab SGLT2i Tacrolimus mTORi (everolimus/sirolimus) Other C3G medication (specify)
Disease management: Duration of C3G treatments during follow-up | Up to 12 months follow-up
  Duration of each of the following C3G treatments during the follow-up:
  ACEi/ARB Corticosteroids Prednisolone Methylprednisolone Cyclophosphamide Complement inhibitors C5 inhibitors (e.g., eculizumab) Other complement inhibitors (specify) Mycophenolate mofetil Rituximab SGLT2i Tacrolimus mTORi (everolimus/sirolimus) Other C3G medication (specify)
Disease management: Number of participants by reason of discontinuation of C3G treatments during follow-up | Up to 12 months follow-up
  treatments during the follow-up: ACEi/ARB Corticosteroids Prednisolone Methylprednisolone Cyclophosphamide Complement inhibitors C5 inhibitors (e.g., eculizumab) Other complement inhibitors (specify) Mycophenolate mofetil Rituximab SGLT2i Tacrolimus mTORi (everolimus/sirolimus) Other C3G medication (specify)
Disease management: Number of participants with antibiotic treatment related to C3G during follow- up | Up to 12 months follow-up
  Any antibiotic therapy during follow-up No Yes
Disease management: Adherence to iptacopan treatment - PDC | Up to 12 months follow-up
  PDC calculated as the total number of days between iptacopan initiation and treatment discontinuation or death. Patients are censored upon disenrollment or reaching the end of follow-up
Disease management: Number of participants by adherence to iptacopan treatment | Up to month 12 follow-up
  PDC < 80% PDC ≥ 80%
Disease management: Number of participants with discontinuation of iptacopan during follow-up | Up to 12 months follow-up
  Number of participants with discontinuation of iptacopan during follow-up and reason for discontinuation of iptacopan
Disease management: Time to iptacopan treatment discontinuation - TTD | Up to 12 months follow-up
  Time from iptacopan initiation to iptacopan discontinuation or death. Patients are censored upon disenrollment or reaching the end of follow-up
Disease management: Number of participants with C3G treatment change after iptacopan discontinuation | Up to 12 months follow-up
  Reason of discontinuation of each of the following C3G treatments during the follow-up:
  ACEi/ARB Corticosteroids Prednisolone Methylprednisolone Cyclophosphamide Complement inhibitors C5 inhibitors (e.g., eculizumab) Other complement inhibitors (specify) Mycophenolate mofetil Rituximab SGLT2i Tacrolimus mTORi (everolimus/sirolimus) Other C3G medication (specify)
Disease management: Numbre of participants by antibiotic treatment related to C3G during follow-up | Up to 12 months follow up
  Any antibiotic therapy during follow-up No Yes
Disease management: Adherence to iptacopan treatment - PDC, % | Up to 12 months follow up
  PDC calculated as the total number of days between iptacopan initiation and treatment discontinuation or death. Patients are censored upon disenrollment or reaching the end of follow-up
Disease management: Adherence to iptacopan treatment, n (%) | Up to 12 months follow up
  PDC < 80% PDC ≥ 80%
Disease management: Number of participants discontinuing iptacopan during follow-up | Up to 12 months follow up
  Discontinuation of iptacopan, with no resumption during the follow-up period. No Yes
Disease management: Number of participants by reason for discontinuation of iptacopan, n (%) | Up to 12 months follow up
  Concerning only patients with iptacopan discontinuation during follow-up. Infection Other adverse effects Death Loss to follow-up Other reasons (to be potentially defined during analysis)
Disease management: Time to iptacopan treatment discontinuation - TTD, days | Up to 12 months follow up
  Time from iptacopan initiation to iptacopan discontinuation or death. Patients are censored upon disenrollment or reaching the end of follow-up
Disease management: C3G treatment change after iptacopan discontinuation, n (%) | Up to 12 months follow up
  Concerning only patients with iptacopan discontinuation during follow-up. No Yes ACEi/ARB Corticosteroids Prednisolone Methylprednisolone Cyclophosphamide Complement inhibitors C5 inhibitors (e.g., eculizumab) Other complement inhibitors (specify) Mycophenolate mofetil Rituximab SGLT2i Tacrolimus mTORi (everolimus/sirolimus) Other C3G medication (specify)
Healthcare resource utilization: Number of hospitalizations during the 12-month period before baseline | Baseline
  Number of hospitalizations, for any cause, during the 12- month period before baseline
Healthcare resource utilization: Number of participants by cause of first hospitalization during the 12-month period before baseline | Baseline
  Concerns only patients with 1 or more hospitalizations during the 12-month period before baseline.
Healthcare resource utilization: Length of first hospitalization during the 12-month period before baseline | Baseline
  Concerns only patients with 1 or more hospitalizations during the 12-month period before baseline
Healthcare resource utilization: Number of participants bu cause of first readmission after first hospitalization during the 12-month period before baseline | Baseline
  Concerning only patients with 2 or more hospitalizations during the 12-month period before baseline
Healthcare resource utilization: Length of first readmission after first hospitalization during the 12-month period before baseline | Baseline
  Concerns only patients with 2 or more hospitalizations during the 12-month period before baseline
Healthcare resource utilization: Number of hospitalizations due to infection during the 12-month period before baseline | Baseline
  Number of hospitalizations due to infection during the 12-month period before baseline by Type (incl. pathogen) of infections
Healthcare resource utilization: Number of hospitalizations during follow-up | Up to 12 months follow-up
  Number of hospitalizations, for any cause, from baseline to 12-month follow-up
Healthcare resource utilization: Number of participants by cause of first hospitalization during follow-up | Up to 12 months follow-up
  Concerns only patients with 1 or more hospitalizations during the follow-up period.
  Categories to be defined at the analysis stage.
Healthcare resource utilization: Length of first hospitalization during follow-up | Up to 12 months follow-up
  Concerns only patients with 1 or more hospitalizations during the follow-up period
Healthcare resource utilization: Number of participants by cause of first readmission after first hospitalization during follow-up | Up to 12 months follow-up
  Concerning only patients with 2 or more hospitalizations during the follow-up period.
  Categories to be defined at the analysis stage.
Healthcare resource utilization: Length of first readmission after first hospitalization during follow-up | Up to 12 months follow-up
  Concerning only patients with 2 or more hospitalizations during the follow-up period
Healthcare resource utilization: Number of hospitalizations due to infection during follow-up | Up to 12 months follow-up
  Number of hospitalizations due to infection during follow-up and Type (incl. pathogen) of infections

CONTACTS AND LOCATIONS:
Overall Officials: Novartis pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No